CLINICAL TRIAL: NCT01848171
Title: Effects of Long-term L-thyroxine Replacement on Serum Lipid and Atherosclerosis in Patients With Hypothyroidism
Brief Title: Effects of L-thyroxine Replacement on Serum Lipid and Atherosclerosis in Hypothyroidism
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Jia-jun Zhao, Professor, Shandong Provincial Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20130328
Record Dates: First submitted 2013-05-02; First posted 2013-05-07 (Estimated); Last update posted 2023-01-18 (Actual); Status verified 2022-05

CONDITIONS: Hypothyroidism; Thyroid Diseases; Endocrine System Diseases
Keywords: Hypothyroidism; Lipid; Atherosclerosis; Oxidative Stress; Chronic Inflammation; Endothelial Function; Adipocytokine; L-thyroxine; coronavirus disease 2019 (COVID-19)
MeSH Terms: conditions — Hypothyroidism; Thyroid Diseases; Endocrine System Diseases; Atherosclerosis; COVID-19 | interventions — Thyroxine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- L-thyroxine (Active Comparator): Oral administration, tablets, starting dose 25 or 50 micrograms once daily, during the follow-up period
  Interventions: Drug: L-thyroxine
- blank (No Intervention): No intervention

INTERVENTIONS:
Drug: L-thyroxine
  Other Names: Euthyrox
  Arms: L-thyroxine

SUMMARY:
Hypothyroidism is a common clinical entity which is often complicated by dyslipidemia. It is also reported increased risk for incidence of atherosclerosis and resulting coronary heart disease(CHD), heart failure(HF) and cardiovascular(CV) death. The effect of L-thyroxine replacement treatment on serum lipid and atherosclerosis is controversial in hypothyroid patients, especially in those with mild or moderate subclinical hypothyroidism. The present study was designed to investigate whether L-thyroxine replacement was effective in improving serum lipid profiles and retarding atherosclerosis progress.

Studies have shown that hypothyroidism increased the risk of COVID-19 composite poor outcomes. This study also aimed to investigate whether L-thyroxine replacement therapy was effective in reducing the incidence and mortality of COVID-19, and in improving the severity of COVID-19 and COVID-19 related complications.

ELIGIBILITY:
Inclusion Criteria:

* 40~75 years old
* Diagnosis of overt or subclinical hypothyroidism in two occasions with a minimum interval period of three months

Exclusion Criteria:

* Pregnant or lactating women
* Severe hepatic or renal dysfunction
* Psychiatric disabilities, acute cardiovascular and cerebrovascular diseases, chronic respiratory diseases, familiar hypercholesterolemia, malignancy, cholelithiasis, pancreatitis, bowel diseases and other disorders influencing lipid and bile acid metabolism
* Taking lipid-lowering agents and other drugs influencing thyroid function, lipid and bile acid metabolism
* Obviously poor compliance.

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 700 (Estimated)
Dates: Start 2013-07; Primary Completion 2023-07 (Estimated); Study Completion 2023-07 (Estimated)

PRIMARY OUTCOMES:
Rate of First cardiovascular disorder (CVD) Events, CVD Mortality and All-cause Mortality | endpoint of the trail

SECONDARY OUTCOMES:
Change in Serum Lipid Levels | baseline, 3 months, 6 months, every 12 months during the following follow-up period until the trial is completed
Change in Thickness of Blood Vessel Wall | baseline, 3 months, 6 months, every 12 months during the following follow-up period until the trial is completed
Change in Oxidative Stress and Chronic Inflammatory Factors Associated with Atherosclerosis | baseline, 3 months, 6 months, every 12 months during the following follow-up period until the trail is completed
Changes in Serum Metabolome and Lipidome | baseline, 3 months, 6 months, every 12 months during the following follow-up period until the trail is completed

OTHER OUTCOMES:
Rate of COVID-19, COVID-19 Mortality, COVID-19 Related Complications and Severity of COVID-19 | Since January, 2023, every 6 months during the following follow-up period until the trail is completed

CONTACTS AND LOCATIONS:
Overall Officials: Zhao jiajun, Study Chair — Shandong Province Hospital
Locations (1):
- Shandong Provincial Hospital, Jinan, Shandong, China

REFERENCES:
- [Derived] Yao Z, Zhao M, Gong Y, Chen W, Wang Q, Fu Y, Guo T, Zhao J, Gao L, Bo T. Relation of Gut Microbes and L-Thyroxine Through Altered Thyroxine Metabolism in Subclinical Hypothyroidism Subjects. Front Cell Infect Microbiol. 2020 Sep 18;10:495. doi: 10.3389/fcimb.2020.00495. eCollection 2020. PMID 33072620
- [Derived] Liu L, Yu Y, Zhao M, Zheng D, Zhang X, Guan Q, Xu C, Gao L, Zhao J, Zhang H. Benefits of Levothyroxine Replacement Therapy on Nonalcoholic Fatty Liver Disease in Subclinical Hypothyroidism Patients. Int J Endocrinol. 2017;2017:5753039. doi: 10.1155/2017/5753039. Epub 2017 Apr 4. PMID 28473851